CLINICAL TRIAL: NCT01482910
Title: A Randomized, Double-masked, Photodynamic Therapy-controlled Phase-3 Study of the Efficacy, Safety, and Tolerability of Intravitreal VEGF Trap-Eye in Chinese Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: VEGF Trap-Eye: Investigation of Efficacy and Safety in Chinese Subjects With Wet AMD (Age-Related Macular Degeneration)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13406
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept; Verteporfin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aflibercept injection (EYLEA, VEGF Trap-Eye, BAY86-5321) (Experimental): Participants received 2.0 mg intravitreal aflibercept injection (IAI) every 4 weeks for the first 12 weeks, followed by additional 2.0 mg IAI every 8 weeks until week 48. Additionally, sham photodynamic therapy (PDT) treatments was administered as needed.
  Interventions: Biological: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- PDT treatments (Active Comparator): Participants received PDT as needed. Additionally, sham IAI injections was administered until week 28. Thereafter, participants received active IAI treatment until week 48.
  Interventions: Drug: Visudyne

INTERVENTIONS:
Biological: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Participants in the VEGF Trap-Eye group received intravitreal injections every 8 weeks following a loading phase with injections given every 4 weeks for an overall treatment period of 48 weeks. Additionally, sham PDT treatments was administered as needed.
  Arms: Aflibercept injection (EYLEA, VEGF Trap-Eye, BAY86-5321)
Drug: Visudyne — Participants in the PDT group (Visudyne group) received Visudyne as needed. Additionally, sham IVT injections was administered until week 28. Thereafter, subjects in the PDT group received active (= no sham) VEGF Trap-Eye treatment until week 48.
  Arms: PDT treatments

SUMMARY:
This study will assess the efficacy and safety of intravitreally (IVT), i.e. directly into the eye administered VEGF Trap-Eye compared with photodynamic therapy (PDT) on visual function in Chinese subjects with age-related neovascular or "wet" age-related macular degeneration.

Subjects will be randomized in a 3:1 ratio to either receive VEGF Trap-Eye or PDT. Both treatment groups will receive the other treatment as a sham procedure.

DETAILED DESCRIPTION:
Adverse events collection will be covered in Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Men and women ≥ 50 years of age.
* Active predominantly classic subfoveal choroidal neovascularization (CNV) lesions secondary to wAMD (wet Age-Related Macular Degeneration)
* BCVA (best corrected visual acuity) of 20/40 to 20/320 in the study eye

Exclusion Criteria:

* Only one functional eye
* Presence of CNV with an origin other than wAMD
* Any prior ocular or systemic treatment or surgery for wAMD, except dietary supplements or vitamins

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- China (10):
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Xi'an, Shaanxi
  - Qingdao, Shandong
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | PDT Treatments
Started | 228 | 76
Completed Week 28 | 216 | 71
Completed | 213 | 67
Not Completed | 15 | 9
Not completed — Adverse Event | 6 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | PDT Treatments | Total
Number analyzed (Participants) | 228 | 76 | 304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (8.8) | 64.9 (8.5) | 65.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 22 | 108
  Male | 142 | 54 | 196

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by ETDRS Letter Score at Week 28 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better functioning.
Time Frame: Baseline and at week 28
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | PDT Treatments
Number analyzed (Participants) | 228 | 76
Letters correctly read | 14.0 (12.1) | 3.9 (14.6)
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs PDT Treatments; Null hypothesis: mean changes are identical in both groups. A sample size of 300 subjects with a 3:1 (EYLEA to PDT) randomization ratio is sufficient to detect the superiority of EYLEA to PDT assuming a two-sided alpha level of 0.05, a power of 90%, a treatment difference of 7.5 letters and a common standard deviation of 14 letters; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing procedure was used in the order of pre-defined fixed sequence (primary endpoint first, then confirmatory secondary efficacy point next). A two-sided significance level of 0.05 was used; ANCOVA with baseline BCVA as a covariate, and treatment group and baseline BCVA group (<45 letters vs ≥45 letters) as fixed factors; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [6.8 to 13.4] — Least square mean difference (EYLEA-PDT) was estimated from ANCOVA, where a positive value is in favor of EYLEA

2. Secondary Outcome: Percentage of Participants Who Lost Fewer Than 15 Letters at Week 28 - LOCF
Description: as for outcome 1
Time Frame: At week 28
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) | PDT Treatments
Number analyzed (Participants) | 228 | 76
Percentage of participants | 98.7 | 92.1
Statistical Analysis 1: Comparison: Aflibercept Injection (EYLEA, VEGF Trap-Eye, BAY86-5321) vs PDT Treatments; Null hypothesis: proportions are identical in both groups; Test type: Superiority or Other; p = 0.0359, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; CMH adjusted for baseline BCVA group (<45 letters vs ≥45 letters); Risk Difference (RD) = 6.6, 95% CI 2-sided [0.4 to 12.9] — Proportion difference (EYLEA-PDT) was estimated from CMH, where a positive value is in favor of EYLEA

ADVERSE EVENTS:
Time Frame: From the first study drug injection until 30 days after the last study drug injection at the latest up to week 52
Groups:
- Aflibercept Injection, up to Week 28: Participants received 2.0 mg intravitreal aflibercept injection (IAI) every 4 weeks for the first 12 weeks, followed by additional 2.0 mg IAI every 8 weeks until week 48. Additionally, sham photodynamic therapy (PDT) treatments was administered as needed. The data up to week 28 was reported.
- PDT Treatments, up to Week 28: Participants received PDT as needed. Additionally, sham IAI injections was administered until week 28. Thereafter, participants received active IAI treatment until week 48. The data up to week 28 was reported.
- Aflibercept Injection, From Week 28 to Week 52: Participants received 2.0 mg intravitreal aflibercept injection (IAI) every 4 weeks for the first 12 weeks, followed by additional 2.0 mg IAI every 8 weeks until week 48. Additionally, sham photodynamic therapy (PDT) treatments was administered as needed. The data from week 28 up to week 52 was reported.
- PDT Then Aflibercept Injection, From Week 28 to Week 52: Participants received PDT as needed. Additionally, sham IAI injections was administered until week 28. Thereafter, participants received active IAI treatment until week 48. The data from week 28 up to week 52 was reported.
Arm/Group | Aflibercept Injection, up to Week 28 | PDT Treatments, up to Week 28 | Aflibercept Injection, From Week 28 to Week 52 | PDT Then Aflibercept Injection, From Week 28 to Week 52
Serious Adverse Events (participants affected / at risk) | 13/228 | 4/76 | 5/216 | 3/71
Other Adverse Events (participants affected / at risk) | 77/228 | 33/76 | 18/216 | 9/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept Injection, up to Week 28 (N=228) | PDT Treatments, up to Week 28 (N=76) | Aflibercept Injection, From Week 28 to Week 52 (N=216) | PDT Then Aflibercept Injection, From Week 28 to Week 52 (N=71)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 2 | 3 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept Injection, up to Week 28 (N=228) | PDT Treatments, up to Week 28 (N=76) | Aflibercept Injection, From Week 28 to Week 52 (N=216) | PDT Then Aflibercept Injection, From Week 28 to Week 52 (N=71)
Conjunctival haemorrhage (Eye disorders) | 14 | 4 | 13 | 4
Retinal haemorrhage (Eye disorders) | 9 | 4 | 0 | 0
Retinal pigment epitheliopathy (Eye disorders) | 12 | 8 | 6 | 1
Visual acuity reduced (Eye disorders) | 16 | 11 | 6 | 5
Subretinal fluid (Eye disorders) | 2 | 4 | 2 | 1
Macular fibrosis (Eye disorders) | 27 | 8 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 4 | 6 | 0
Intraocular pressure increased (Investigations) | 12 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less